CLINICAL TRIAL: NCT01897064
Title: The Influence of Aerobic Exercise on Cognitive Functioning in Schizophrenia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6508; R21 096132 (Other Grant/Funding Number: NIMH)
Record Dates: First submitted 2013-06-26; First posted 2013-07-11 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Cognition; Aerobic Exercise
MeSH Terms: conditions — Schizophrenia | interventions — Exercise; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aerobic Exercise (Experimental): Up to 36 sessions of aerobic exercise (12 weeks of 3 times/week, 60-minute exercise sessions) in small groups (3-5 individuals), in addition to standard psychiatric treatment.
  Interventions: Behavioral: Aerobic Exercise
- Standard Psychiatric Treatment (Active Comparator): 12 weeks of standard psychiatric treatment.
  Interventions: Other: Standard Psychiatric Treatment

INTERVENTIONS:
Behavioral: Aerobic Exercise — 36 sessions of aerobic exercise (12 weeks of 3 times/week, 60-minute exercise sessions) in small groups (3-5 individuals), in addition to standard psychiatric care.
  Other Names: AE
  Arms: Aerobic Exercise
Other: Standard Psychiatric Treatment — Standard psychiatric treatment.
  Other Names: Treatment As Usual (TAU)
  Arms: Standard Psychiatric Treatment

SUMMARY:
The aim of this study is to look at the effects of Aerobic Exercise (AE) on daily and neurocognitive functioning including memory, attention, the ability to plan activities, and learn new information. Participants will be assigned by chance to receive regular care or exercise sessions in addition to regular care. This study will allow determining the potential positive influence of AE on cognitive and daily functioning in individuals with schizophrenia.

DETAILED DESCRIPTION:
Individuals with schizophrenia often display cognitive difficulties. Studies among non-clinical populations suggest that Aerobic Exercise (AE) training is effective in increasing both aerobic fitness and cognitive functioning. However, these associations have not been studied among individuals with schizophrenia, despite the presence of highly sedentary lifestyle in this population To elucidate this putative link, the present study will evaluate the influence of AE on cognitive functioning and daily functioning in individuals with schizophrenia using a single-blind, randomized clinical trial. Outpatient individuals with schizophrenia receiving treatment will be randomly assigned to AE training or Treatment As Usual (TAU). Participants in the AE training will undergo a 12-week, 3 times per week, 1-hour AE sessions. All participants will continue their regular psychiatric and medical care. Assessments of neurocognitive and daily functioning abilities, along with symptom severity, and physiological and behavioral measures of aerobic fitness will be completed before and after the 12-week program.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between ages 18-55.
* Have capacity to give informed consent.
* English speaking.
* Have a DSM-IV diagnosis of schizophrenia.
* Taking antipsychotic medication for at least 8 weeks and on current doses for 4 weeks, and/or injectable depot antipsychotics with no change in last 3 months.
* Medically cleared to exercise.

Exclusion Criteria:

* Lacks capacity to give informed consent.
* Have used street drugs within the past 4 weeks.
* Have history of of hypertension of cardiac conditions.
* Have history of active suicidal ideation or serious self-destructive behavior.
* Have history of violence or aggressive behavior.
* Have history of neurological or medical conditions known to seriously affect the brain.
* Pregnant or nursing.
* Completing more than 2 hours of moderate or higher levels of aerobic exercise per week.
* Participation in a study of cognition during the previous 2 months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2012-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in MATRICS Consensus Cognitive Battery scores at 12 weeks | Baseline and after 12 weeks.
  Standardized battery designed to measure cognition specifically in individuals in schizophrenia.
Change from Baseline in VO2Max (maximal oxygen consumption) at 12 weeks | Baseline and after 12 weeks
  The VO2Max (maximal oxygen consumption) test measures maximum ability to consume oxygen and is a key indicator of aerobic fitness.
Change from Baseline in 6-Minute Walk Test (6MWT) score at 12 weeks | Baseline and after 12 weeks
  The six-minute walk test (6MWT) measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes.
Change from Baseline in Daily Functioning Assessments at 12 weeks | Baseline and after 12 weeks
  Measures include: The Specific Levels of Functioning Scale (SLOF), Quality of Life Scale (QLS), and Quality of Life Scale (QoL-16).

SECONDARY OUTCOMES:
Change from Baseline in The Cognitive Neuroscience Treatment Research to Improve Cognition in Schizophrenia program (CNTRICS) measures at 12 weeks | Baseline and after 12 weeks
  Measures include: AX-CPT/Dot Pattern Expectancy (DPX) Task, Recent Probe Task, Relational Item Specific Encoding Task, Probabilistic Reward Task, Sustained Attention Task with and without Distraction, Automated Operation Span Task (OSPAN), and Automated Symmetry Span Task (SSPAN).

CONTACTS AND LOCATIONS:
Overall Officials: David Kimhy, Ph.D., Principal Investigator — Columbia University & New York State Psyciatric Institute
Locations (1):
- Columbia University & New York State Psyciatric Institute, New York, New York, United States

REFERENCES:
- [Derived] Kimhy D, Khan S, Ayanrouh L, Chang RW, Hansen MC, Lister A, Ballon JS, Vakhrusheva J, Armstrong HF, Bartels MN, Sloan RP. Use of Active-Play Video Games to Enhance Aerobic Fitness in Schizophrenia: Feasibility, Safety, and Adherence. Psychiatr Serv. 2016 Feb;67(2):240-3. doi: 10.1176/appi.ps.201400523. Epub 2015 Oct 1. PMID 26423100